CLINICAL TRIAL: NCT05373056
Title: Effects of Scapular Strength Exercise for Patients With Lateral Epicondylalgia a Randomized Clinical Trial
Brief Title: Effects of Scapular Strength Exercise for Patients With Lateral Epicondylalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alejandro Ayuso Pablo, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAMaster123
Record Dates: First submitted 2022-05-03; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylalgia; tennis elbow; lateral epicondylitis; exercise; scapular muscle
MeSH Terms: conditions — Tennis Elbow; Motor Activity

STUDY DESIGN:
Intervention Model Description: There are two groups, the control group and the experimental group. In the control group, only the conventional exercise program for epicondylar muscles will be performed and the experimental group will also perform a scapular exercise program. Group assignment is randomized using the G* POWER software program.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Control group (Active Comparator): They will performer the conventional exercise program por epicondylar muscles.
  Interventions: Behavioral: Conventional program
- Group 2 - Experimental group (Experimental): The experimental group will perform the conventional exercise program and also a scapular exercise program.
  Interventions: Behavioral: Scapular program

INTERVENTIONS:
Behavioral: Scapular program — the patient will be in prone. With the elbow extended, begin by raising the shoulder above the head, keeping the upper extremity in line with the fibers of the lower trapezius. The participant will then remain pronated with the elbow flexed at 90 degrees and the shoulder abducted and externally rotated. Starting from this position, you should exert the force towards external rotation and then return to internal rotation. For the last exercise, the subject will be placed in a standing position holding the elastic band with one hand while the other end will fix it to the ground, while stepping on it with the foot. You will start the movement with a shoulder elevation in the plane of the scapula above 120 degrees and then perform the eccentric returning to the starting position.
  Arms: Group 2 - Experimental group
Behavioral: Conventional program — They will be performing a combination of concentric-eccentric type contractions adding an isometric contraction
  Arms: Group 1- Control group

SUMMARY:
the aim of the study is to determine whether a scapular strength exercise program combined with a conventional exercise program in epicondylar region in patients with lateral epicondylalgia produces statistically significant improvements in pain in the short and medium term compared to a conventional exercise program.

DETAILED DESCRIPTION:
It is a single-blind clinical trial design, with third-party evaluation. There are two groups, the control group and the experimental group. In the control group, only the conventional exercise program for epicondylar muscles will be performed and the experimental group will also perform a scapular exercise program. Group assignment is randomized using the G* POWER software program, following the inclusion and exclusion criteria. Variables related to pain, functionality, pressure pain threshold, prehensile strength and quality of life will be measured. The study will last 7 months.

ELIGIBILITY:
Inclusion Criteria:

* tenderness over the epicondyle.
* Clinical diagnosis of LD for at least 3 months.
* Positive Mills and Maudsley test

Exclusion Criteria:

* Patients with carpal tunnel syndrome, rheumatoid arthritis, cervical root syndrome, rotator cuff tendinopathy.
* Fractures or surgical history in the shoulder or elbow.
* History of elbow immobilization.
* Limitation in range of motion of the shoulder.
* Having undergone upper limb surgery in the last 6 months
* Unhealed wound in the region in the treatment area
* Impairment at a cognitive level that makes understanding with the therapist impossible.
* Neural entrapment of the radial nerve.
* Corticosteroid infiltration in the upper limb to be treated.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale for Pain | 4 weeks
  It will be measured with a 10 cm long horizontal line with descriptors at each end to help subjects identify their level of pain. The participants will mark with a cross the point of the line that most corresponds to the intensity of their symptoms. When interpreting the VAS, the respondent's cross position is usually assigned a score between 0 and 10. If documented on paper, pressures can simply be transferred to a scale of 100 values using a millimeter tape measure, although division into hundredths is considered sensitive enough.

SECONDARY OUTCOMES:
Functionality | 4 weeks
  measured with "the patient-rated tennis elbow evaluation Questionnaire".It is made up of 15 items, 5 focused on pain and the other 10 distributed between activities of daily living (4 items) and more specific activities (6 items). The result of each item is represented on a scale from 0 (totally painless activity) to 10 (maximum pain imaginable), so the total score can vary between 0 and 150.
grip strength | 4 weeks
  measured by dynamometer
The Quality of the lifestyle | 4 weeks
  measured with "The Short Form-36 Health Survey Questionnaire".It is evaluated on a scale from 0 to 100, with the highest score being the maximum possible health and well-being. Finally, a total score is obtained from the questionnaire considering a score of 0-19 = very low, 20-39 = relatively low, 40-59 = average, 60-79 = relatively high and 80-100 = very high.
pressure threshold | 4 weeks
  measured by pressure algometer

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro AY Ayuso Pablo, Msc, Principal Investigator — Alcala University
Locations (1):
- Alcala University, Madrid, Alcala de Henares, Spain

IPD SHARING:
Plan to Share IPD: No